CLINICAL TRIAL: NCT02733458
Title: The Efficacy and Safety of Gemcitabine, Etoposide, Dexamethasone and Pegaspargase Chemotherapy (GELAD) With Sandwiched Radiotherapy in the Treatment of Stage IE/II Natural Killer/T-Cell Lymphoma: A Multicenter, Prospective Study
Brief Title: GELAD Chemotherapy and Sandwiched Radiotherapy in the Treatment of Stage IE/IIE Natural Killer/T-cell Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Rong Tao, Dr, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1601
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gemcitabine; Etoposide; Dexamethasone; pegaspargase; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GELAD/Radiation (Experimental): Patients will be initially treated with two cycles GELAD chemotherapy, followed by 50-56Gy radiotherapy, and completed with another two cycles GELAD chemotherapy. GELAD chemotherapy will be repeated every 21 days. Radiotherapy will be delivered in 25-32 fractions.
  Interventions: Drug: GELAD; Radiation: Radiotherapy

INTERVENTIONS:
Drug: GELAD — Gemcitabine, 1.0g/m2/d IV, day 1 Etoposide, 60mg/m2 IV, day 1 to day 3 Dexamethasone, 40mg/d IV, day 1 to day 4 Pegaspargase, 2000IU/m2/d IM, day 4
  Other Names: Gemcitabine, Etoposide, Dexamethasone, Pegaspargase
Radiation: Radiotherapy — Radiotherapy: 50-56Gy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of gemcitabine, etoposide, pegaspargase and dexamethasone (GELAD) chemotherapy and sandwiched radiotherapy as first-line treatment in patients with de novo stage IE/IIE extranodal natural killer/T-cell lymphoma, nasal type.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTCL), nasal type, is a rare subtype of non-Hodgkin lymphoma (NHL) with relatively high incidence in China. Radiotherapy alone for stage IE/IIE diseases has good response rate but with high relapse rates, ranging from 20-50%. The combination of chemotherapy and radiotherapy improved the long-term survival for patients with stage IE/IIE diseases. But the optimal treatment schedule has not been established. This study is designed with two cycles GELAD chemotherapy, followed by 50-56Gy radiotherapy, and completed with additional two cycles GELAD chemotherapy. The efficacy and safety of this sandwiched chemoradiotherapy in the treatment of stage IE/IIE ENKTCL will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of extranodal natural killer/T-cell lymphoma, nasal type, previously untreated
* Eastern Cooperative Oncology Group (ECOG ) performance status 0~3
* Stage IE to IIE disease with at least one measurable lesion in the nasal cavity, paranasal sinuses, orbit, pharynx, Waldeyer's ring, or oral cavity.
* Preserved organ functions for: absolute neutrophil counter (ANC)>1.0×109/L, Platelet>50×109/L, hemoglobin>80g/L, total bilirubin (TBIL)<2×ULN, alanine transaminase (ALT)<2×ULN, serum creatinine<1.5×ULN，fibrinogen≥1.0g/L, LVEF≥50%
* No history of chemotherapy or radiotherapy.
* Signed Informed consented

Exclusion Criteria:

* Concurrent cancers need surgery or chemotherapy within 6 months.
* Significant complications: LVEF≤50%, coagulopathy, autoimmune disease, severe infection, or liver cirrhosis, hemophagocytic lymphohistiocytosis.
* Mental disorders.
* Pregnant or lactation
* HIV, hepatitis virus C (HCV), or active hepatitis virus B (HBV) infection with HBV DNA≥105 copies/ml.
* History of pancreatitis
* Known history for grade 3/4 allergy to the drugs in chemotherapy regimen.
* Enrolled in other trial treatment

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 28 days after 4 cycles of chemotherapy
  The complete response rate will be assessed on day 28 after the 4th course of chemotherapy.

SECONDARY OUTCOMES:
Progression free survival | 2-year
  Progression free survival is the time from entry onto the treatment until lymphoma progression or death of any reason.
Overall Response rate | 28 days after 4 cycles of chemotherapy
  The complete response rate will be assessed on day 28 after the 4th course of chemotherapy.
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course and then every 3 months for 2 years
  Treatment-Related Adverse Events will be assessed and graded by NCI CTCAE v4.0.
Overall survival | 2-year
  Overall survival is defiend as the time from entry onto the treatment until death of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Xinhua hospital, Shanghai Jiao Tong University of Medicine
Locations (7):
- China (7):
  - Shanghai Dong Fang hospital, Shanghai, Shanghai Municipality
  - Department of Hematology, Renji Hospital, Shanghai, Shanghai Municipality
  - South Renji hospital, Shanghai, Shanghai Municipality
  - Xin Jiang People's Hospital, Ürümqi, Xinjiang
  - Shanghai Ninth Peoples' Hospital, Shanghai
  - Shanghai Eye and ENT Hospital of Fudan University, Shanghai
  - Xinhua Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Y, Tian S, Xu L, Ma Y, Zhang W, Wang L, Jin L, Liu C, Zhu C, Li Z, Hao S, Zhong H, Ding H, Tao R. GELAD chemotherapy with sandwiched radiotherapy for patients with newly diagnosed stage IE/IIE natural killer/T-cell lymphoma: a prospective multicentre study. Br J Haematol. 2022 Feb;196(4):939-946. doi: 10.1111/bjh.17960. Epub 2021 Nov 21. PMID 34806163